CLINICAL TRIAL: NCT00431288
Title: Efficacy of a Nutrition Intervention Emphasizing Fruits, Vegetables and Dairy to Lower Blood Pressure in Adolescents
Brief Title: A Nutrition Intervention to Lower Blood Pressure in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sarah C. Couch, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHA 0355332B
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: nutrition; adolescent nutrition; blood pressure; hypertension; diet therapy; patient education
MeSH Terms: conditions — Hypertension | interventions — Fruit; Vegetables

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All measurements were made in the Cincinnati Children's Hypertension Clinic by trained clinic staff blinded to treatment assignment.

ARMS (2):
- DASH intervention (Experimental): The DASH diet used in this intervention was slightly modified from the original version of the DASH diet for adults to more closely conform to the unique nutritional needs of adolescents. Details of the intervention have been published (Couch, SC et al. J Pediatrics 2008; 152: 494-501)
  Interventions: Behavioral: diet high in fruits, vegetables, and dairy
- Routine Care (Other): Routine care did not deviate from the nutrition counseling that was routinely given to all new patients at the Cincinnati Children's Hypertension Clinic. Details of routine care have been published (Couch, SC et al. J Pediatrics 2008; 152: 494-501)
  Interventions: Other: Routine nutrition care

INTERVENTIONS:
Behavioral: diet high in fruits, vegetables, and dairy
  Other Names: DASH dietary pattern
  Arms: DASH intervention
Other: Routine nutrition care
  Other Names: Routine Care
  Arms: Routine Care

SUMMARY:
The purpose of this study is to evaluate the efficacy of a 12-week, clinic-based, behavioral nutrition intervention emphasizing fruits, vegetables, and low fat dairy compared to routine nutrition care on changing diet quality and blood pressure post-treatment and at short-term follow-up in adolescents with hypertension.

DETAILED DESCRIPTION:
Among youth, hypertension is no longer a rare disease, affecting about 7 million children and adolescents. Numbers are increasing with the evolving pediatric obesity epidemic in the US. More adolescents than children have primary hypertension, which tracks into adulthood and has been linked with preclinical indicators of adverse cardiovascular events in adults. Early prevention and intervention efforts are needed to address this increasing public and individual health problem. The purpose of this project is to evaluate the immediate and sustained impact of a 3-month clinic-based behavioral nutrition intervention emphasizing a diet high in fruits, vegetables, and low fat dairy, and low in fat and sodium (the DASH intervention) versus routine nutrition care on changing diet quality and blood pressure in adolescents with pre-hypertension or hypertension. The DASH intervention will include a printed participant manual, 1 individual counseling session with a dietitian, 4 mailings and 10 telephone calls on behavioral strategies to promote dietary change. Routine care will include 1 individual counseling session with a dietitian on dietary guidelines consistent with those of the National High Blood Pressure Education Program. Adolescents with prehypertension or hypertension will be randomly assigned to the DASH intervention or routine nutrition care after pre-treatment assessment. Post-treatment and at 3-month follow-up, outcome measures will be assessed including dietary intake and blood pressure. Our expectations are that the DASH intervention will significantly improve dietary quality and blood pressure in adolescents with elevated blood pressure compared to that observed as a result of routine nutrition care. The findings from this study are expected to improve the manner in which hypertension among adolescents is being treated in the clinical setting and contribute to the enhancement of the cardiovascular health of the target population.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of prehypertension or stage 1 hypertension
* age 11-18 years
* english speaking

Exclusion Criteria:

* stage 2 or secondary hypertension
* target organ damage or symptomatic hypertension
* type 1 or 2 diabetes
* treated with anti-hypertensive medications or other blood pressure altering medications
* are unwilling to stop use of vitamins, minerals or antacids containing calcium or magnesium
* do not have full medical clearance from a physician to participate

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | change from baseline BP at immediately post-treatment (3 months)
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurements were performed with a mercury sphygmomanometer according to standardized procedures. SBP and DBP were measured two times and averaged. SBP and DBP z-scores were determined from these average measurements based on established norms.

SECONDARY OUTCOMES:
Diet quality Indicators | change from baseline diet quality indicators at immediately post-treatment (3 months)
  Dietary intake was assessed with 3, 24-hour recalls collected over a 2-week period (2 weekdays and 1 weekend day) before each assessment visit using the validated multi-pass method. Recalls were collected from the adolescent by telephone interview and coded by a trained research dietitian. Adolescents were trained in the use of a 2-dimensional food portion size model to enhance recall of different food volumes and dimensions. Food recalls were analyzed for selected nutrients and servings of fruits, vegetables, low fat dairy foods and high sodium and fat containing foods using the Minnesota Nutrient Data Systems software (version 5.0, 2003). Indicators of diet quality were recorded as average number of daily servings of fruits, vegetables, low fat dairy foods and high fat and sodium containing foods.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Couch, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Couch SC, Saelens BE, Levin L, Dart K, Falciglia G, Daniels SR. The efficacy of a clinic-based behavioral nutrition intervention emphasizing a DASH-type diet for adolescents with elevated blood pressure. J Pediatr. 2008 Apr;152(4):494-501. doi: 10.1016/j.jpeds.2007.09.022. Epub 2007 Nov 5. PMID 18346503